CLINICAL TRIAL: NCT06974084
Title: A Multi-Center Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy of Maraviroc and Atorvastatin for the Treatment of Subjects With Long COVID/Post-Acute Sequalae of Covid (PASC)
Brief Title: Investigating Measurable PRO Acuity Trial (IMPACT) is a Multi-Center Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy of Maraviroc and Atorvastatin to Improve Neurocognitive and Physical Function of Subjects With Long COVID-19/Post-Acute Sequelae of COVID-19 (PASC).
Acronym: IMPACT-LC
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: HealthBio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IMPACT Long Covid Treatment
Record Dates: First submitted 2025-05-07; First posted 2025-05-15 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Long COVID
Keywords: Long Covid; Post-COVID syndrome (PCS)
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome | interventions — Maraviroc; Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Study Drug; Combination of Maraviroc (300mg) and Atorvastatin (10mg) given twice daily (Active Comparator): Subjects randomized to maraviroc/atorvastatin will receive maraviroc 300 mg and atorvastatin 10 mg twice daily oral for 16 weeks.
  Interventions: Drug: Maraviroc (MVC); Drug: Atorvastatin, 10mg, 20mg, 40mg
- Placebo of Maraviroc (300mg) and Atorvastatin (10mg) given twice daily (Placebo Comparator)
  Interventions: Drug: Placebo, Maraviroc; Drug: Placebo, Atorvastatin

INTERVENTIONS:
Drug: Maraviroc (MVC) — Maraviroc, 300mg per tablet. Atorvastatin, 10mg per tablet
  Arms: Study Drug; Combination of Maraviroc (300mg) and Atorvastatin (10mg) given twice daily
Drug: Atorvastatin, 10mg, 20mg, 40mg — Atorvastatin, 10mg will be given twice daily oral along with Maraviroc, 300-mg
  Arms: Study Drug; Combination of Maraviroc (300mg) and Atorvastatin (10mg) given twice daily
Drug: Placebo, Maraviroc — Placebo of Maraviroc, 300mg
  Arms: Placebo of Maraviroc (300mg) and Atorvastatin (10mg) given twice daily
Drug: Placebo, Atorvastatin — Placebo of Atorvastin, 10mg
  Arms: Placebo of Maraviroc (300mg) and Atorvastatin (10mg) given twice daily

SUMMARY:
The IMPACT Long Covid Treatment clinical study (IMPACT-LC) is testing two repurposed and previously approved drugs, Maraviroc and Atorvastatin, for the treatment of non-hospitalized subjects with long COVID/Post-Acute Sequelae of COVID (PASC). The main goals of the clinical study are to determine if this combination drug therapy can improve neurocognitive and physical functions in Long Covid patients, such as fatigue severity, heart rate, blood pressure, digestion, breathing, dizziness, and cognitive function. A secondary goal is to determine if biomarker levels, measured by a diagnostic test, can improve during treatment. To qualify for the trial, a subject must be an adult ≥ 18 and ≤ 65 years of age and meets the WHO-defined post-COVID-19 condition and has one or more new-onset Long Covid symptom that persist ≥ 6 months after the diagnosis of acute COVID-19 infection. A total of 252 participants will take either two daily doses of two existing medications (Maraviroc and Atorvastatin together as separate tablets) or a placebo (pills with no active ingredient) for 16 weeks. Although these medications are not yet approved for Long Covid, they are FDA-approved for use in treating other health conditions.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 and ≤ 65 years of age at the time of consent
2. Meets WHO-defined post-COVID-19 condition (WHO definition: 'Post COVID-19 condition occurs in individuals with a history of probable or confirmed SARS-CoV-2 infection, usually 3 months from the onset of COVID-19 with symptoms that last for at least 2 months. Common symptoms include fatigue, shortness of breath, cognitive dysfunction but also others and generally have an impact on everyday functioning. Symptoms may be new onset following initial recovery from an acute COVID-19 episode or persist from the initial illness. Symptoms may also fluctuate or relapse over time).
3. One or more new onset symptoms that persisted greater than 6 months after the diagnosis of acute COVID-19 infection. These symptoms include: cognitive impairment (brain fog), migraines, post exertional malaise (PEM), myalgias, arthralgias, severe fatigue, tachyarrhythmias, postural orthostatic tachycardia syndrome (POTS), and shortness of breath.
4. Documented confirmation of previous COVID-19 infection from a positive PCR laboratory test and/or medical records from healthcare provider that coincides with the diagnosis of Long-COVID/PASC.
5. Lyme screen (Borrelia, Bartonella, Babesia) two-tier serologic negative (centrally assessed).
6. Epstein-Barr Virus (EBV) DNA negative (centrally assessed).
7. A long hauler index (LHI) of >0.5
8. FSS score ≥ 36
9. Female participants should be surgically sterilized or post-menopausal or must agree to take effective contraceptive measures during the study period. Adequate methods of birth control include: condoms, male or female, with or without a spermicide; diaphragm or cervical cap with spermicide; intrauterine device; any of the methods that require a prescription (such as contraceptive pills or path) or a male partner who has previously undergone vasectomy.
10. Participant is willing and able to participate in the study and comply with all study requirements.
11. Participant provided signed and dated IRB approved informed consent prior to initiation of any study procedures.

Exclusion Criteria:

1. Participation in another therapeutic clinical trial in the past 2 months.
2. History of allergy or anaphylaxis or allergic reaction to any component of atorvastatin and/or maraviroc.
3. Pre-COVID history of autoimmune conditions, migraines, neuropathy, inflammatory bowel disease (IBD), obsessive-compulsive disorder (OCD), chronic fatigue syndrome, or fatigue duration for ≥5 year, EBV infection, Lyme disease, fibromyalgia, arthritis, chronic obstructive pulmonary disease (COPD), asthma, chronic kidney disease, chronic heart failure (CHF), arrhythmias, bleeding disorders, and anticoagulation therapy.
4. Presence of other conditions or differential diagnosis better explaining the symptoms of the patient than the suspected long COVID/PASC.
5. Hepatic impairment defined as Childs-Pugh Score B or greater.
6. Active/acute infectious diseases like tuberculosis, human immunodeficiency virus infection (HIV), cytomegalovirus (CMV), Lyme, EBV, hepatitis B virus (HBV), hepatitis C virus (HCV).
7. Ongoing immunosuppressive therapy.
8. Use of statins within 6 months of randomization.
9. Concomitant use of cyclosporine, gemfibrozil, tipranavir plus ritonavir, or glecaprevir plus pibrentasvir, or lipid modifying doses (>1 gram/day) of niacin.
10. Severe renal impairment defined as GFR<30.
11. AST:ALT ratio>1.5
12. Elevations in IL-8 (>21 (pg/ml) and or IL-13 (>6.1 pg/ml) (centrally assessed)
13. Pregnant, breastfeeding, or unwilling to practice birth control during participation in the study.
14. History of illicit drug abuse (including marijuana or alcohol abuse) within 3 months of enrollment.
15. Inability to provide consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Fatigue | FSS scores will be taken during screening (0-28 days before the first baseline)at visit 3 (week 8 +/-3D) and at the EOT visit, week 16. The PGI-S score will be collected at Visit One, Day 1, Visit 3 (week 8) and EOT (week 16)
  Two Patient Reported Outcomes for fatigue will be measured: 1)Fatigue Severity Scale (FSS) is a 9-item scale which measures the severity of fatigue and its effect on a person's activities and lifestyle. Each of the nine item about fatigue from the FSS is scored on a Likert scale on which 7 is Strongly Agree and 1 is Strongly Disagree. The total score ranges from 9 to 63, with higher scores indicating greater fatigue severity. A total score of <36 indicates a subject is not suffering from fatigue.
  2)Subjects will be asked to complete the single-item PGI-S (Patient Global Impression of Severity). PGI-S is a single item scale for assessing fatigue severity containing 6 response options from 0 (not present) to 5 (very severe). A one-point change in PGI-S from baseline would represent a minimal individual change that is meaningful.

SECONDARY OUTCOMES:
Improvement in dysautonomia symptoms as reflected by the Composite Autonomic Symptom Score (COMPASS-31) | Scores will be determined at Visit 1 (Day 1), Visit 3 (week-8) and EOT (week -16)
  Difference in the mean Composite Autonomic Symptom Score (COMPASS-31) score at week 8 and week 16 between maraviroc/atorvastatin and placebo.
Improvement in Dyspnea | MRC (Medical Research Council) Dyspnea Scale will be measured at Visit 1 (Day-1), Visit 3 (week-8) and EOT (week-16)
  Difference in mean Medical Research Council (MRC) Dyspnea grade at week 8 and week 16 between maraviroc/atorvastatin and placebo.
Improved Cognitive Function, measured by the PROMIS (Patient-Reported Outcomes Measurement Information System) Cognitive Function v.2.0 - Short Form 6a | Difference in T-score measured at Visit 1 (Day 1), Visit 3 (week-8) and EOT (week-16)
  The PROMIS (Patient-Reported Outcomes Measurement Information System) Cognitive Function v.2.0 - Short Form 6a is a 6-item sub-set scale of the PROMIS Cognitive Function item bank that assesses patient-perceived cognitive deficits. Each item has five response options ranging in value from one to five. The total raw score for a short form with all questions answered, is the sum of the values of the response to each question and ranges between 6 and 30. The raw score is translated in a T-score, a standardized score with a mean of 50 and a standard deviation (SD) of 10.
To assess if maraviroc and atorvastatin decrease the Long Hauler Index (LHI) from baseline to week 8 and from baseline to week 16. | LHI will be measured at Visit 1 (Day-1), Visit 3 (week-8) and EOT (week-16)
  The LHI was developed using machine learning, and built on a tailored panel of cytokines and chemokines specific for abnormalities in cytokine storm conditions and in chronic COVID-19 patients. It generates a severity score spanning the spectrum of disease severity from mild to critical.
To assess the effect of maraviroc and atorvastatin on IncellKINE biomarker levels | IncellKINE test will be run at Visit 1 (Day-1), Visit 3 (week-8) and EOT (week-16)
  Change in mean biomarker levels as measured by the IncellKINE assay from baseline to week 8 and from baseline to week 16.
To determine the safety profile of maraviroc and atorvastatin in patients treated for Long COVID-19 | Adverse event collection will be done during every Visit (Day-1, Week-4, Week-8, Week-12, Week-16 (EOT) and EOS (28-42 Days after last dose)
  Participants report data will be compiled as follows:
  Percentage of participants reporting AEs from Dose 1 to 28 days after the last dose.
  Percentage of participants reporting SAEs from Dose 1 to 28 days after the last dose.
  Percentage of participants reporting AEs leading to discontinuation. Percentage of participants reporting SAEs leading to discontinuation.
To evaluate the PK (pharmacokinetic) profiles of atorvastatin and maraviroc in participants treated for Long COVID-19 | PK reports will be generated from patient samples at Visit 1(Day-1) and Visit 2 (week-4). At any reported SAE, PK profile will also be run.
  Blood samples will be collected from participants receiving 4 weeks of study intervention - samples collected at Visit 1 and 2 - with PK profiles run.
  The PK profiles of atorvastatin and maraviroc will also be measured for all reporting SAE's.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Arizona, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: Undecided